CLINICAL TRIAL: NCT01804985
Title: A Trial of De-escalation and Stopping Treatment in Chronic Myeloid Leukaemia Patients With Excellent Responses to Tyrosine Kinase Inhibitor Therapy
Brief Title: De- Escalation and Stopping Treatment of Imatinib, Nilotinib or sprYcel in Chronic Myeloid Leukaemia
Acronym: DESTINY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Liverpool (Other)
Collaborators: Newcastle University (Other); Imperial College London (Other); University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4203
Record Dates: First submitted 2013-03-03; First posted 2013-03-05 (Estimated); Last update posted 2025-03-14 (Actual); Status verified 2018-09

CONDITIONS: Chronic Myeloid Leukaemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate; nilotinib; Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- De-escalated Treatment (Experimental): Imatinib, nilotinib or dasatinib; de-escalated to half the standard dose for 12 months
  Interventions: Drug: Imatinib; Drug: nilotinib; Drug: dasatinib

INTERVENTIONS:
Drug: Imatinib — Imatinib, nilotinib or dasatinib; de-escalated to half the standard dose for 12 months. If on imatinib, the dose should be decreased to 200mg daily;
  Other Names: Glivec or Gleevec
Drug: nilotinib — Imatinib, nilotinib or dasatinib; de-escalated to half the standard dose for 12 months. if on nilotinib to 200mg twice daily (which is half the standard dose for second line use, since it is anticipated that the vast majority of nilotinib entrants will be receiving 400mg twice daily because of prior imatinib intolerance);
  Other Names: Tasigna
Drug: dasatinib — Imatinib, nilotinib or dasatinib; de-escalated to half the standard dose for 12 months. If on dasatinib then to 50 mg daily.
  Other Names: Sprycel

SUMMARY:
The purpose of this study is to investigate whether some patients with excellent responses to chronic myeloid leukaemia (CML) treatment are being overtreated, and can remain well on either a lower dose of treatment or without treatment at all. The dose of imatinib (Glivec), nilotinib (Tasigna) or dasatinib (Sprycel) treatment will initially be cut to half the standard dose for 12 months, and then treatment will be stopped completely for a further two years. The trial information will also help to develop a de-escalation and stopping strategy for future newly diagnosed CML patients in the next British national CML study (to be known as SPIRIT3).

DETAILED DESCRIPTION:
The next definitive United Kingdom (UK) phase III trial in chronic myeloid leukaemia (CML) will be SPIRIT3, which will open shortly. This will incorporate a de-escalation and stopping strategy for patients who achieve excellent responses after at least 3 years of treatment with a tyrosine kinase inhibitor (TKI).

DESTINY is to act as a pilot for this strategy in SPIRIT3, by defining the proportion of patients that relapse during 12 months of TKI de-escalation followed by 24 months of cessation. DESTINY also includes scientific bolt-on studies, quality of life assessments and health economic evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. CML in first chronic phase.
2. Demonstration of BCR-ABL1 positivity at/shortly after original diagnosis.
3. Written Informed Consent
4. Must have received TKI treatment for at least 3 years.
5. At least 3 molecular results over the preceding 12 months, that fit either of the following groups (results from any UK lab are acceptable):

   * (MR4 group) all the available BCR-ABL1 molecular results over the preceding 12 months are in MR4 (MR4 is defined as a BCR-ABL1/ABL1 ratio of zero, (reported to International Standards (IS) where possible; with at least 10,000 ABL1 control transcripts).
   * (MMR group) some or all BCR-ABL1 molecular results are in major molecular response (MMR), defined here as a BCR-ABL1/ABL1 ratio of 0.1% or less, (reported to International Standard (IS) where possible), but not zero, with at least 10,000 ABL1 control transcripts. If the results over the preceding 12 months are a mix of MMR and undetectable BCR-ABL1, then the patient is eligible for the MMR but not the MR4 group.

Exclusion Criteria:

1. Age under 18
2. Life expectancy predicted to be less than 37 months because of intercurrent illness
3. Presence of serious concomitant illness (e.g. heart, renal, respiratory or active malignant disease) that might preclude completion of the trial
4. CML in accelerated phase or blast crisis at any time
5. Any molecular result during the preceding 12 months that is not in either MMR or MR4.
6. Patients who switched previous licensed TKI treatment (imatinib, nilotinib or dasatinib) twice or more because of intolerance
7. Treatment with higher than standard TKI doses ('standard' is defined as imatinib 400mg daily, nilotinib 400mg twice daily or dasatinib 100mg daily). However, an exception is made for patients who at original diagnosis commenced on either 800mg of imatinib on the SPIRIT1 study, or 140mg (or 70mg b.d) of dasatinib in the Bristol-Myers Squibb 034 study. In each case these latter patients ARE eligible provided they fulfil other molecular criteria, since they do not demonstrate resistant disease.
8. Patients who switched previous licensed TKI treatment (imatinib, nilotinib or dasatinib) because of resistance. Patients treated with lower (but at least 50%) than the standard TKI doses (as defined in previous criterion) for tolerance reasons may be included, but will de-escalate to the same doses as for standard dose patients and will be analysed separately, as they could be seen as undertreated.
9. Previous treatment with ponatinib or bosutinib. Patients who received interferon prior to commencing TKI (even if resistant to their interferon) are eligible, provided their response to TKI fits the entry criteria.
10. Pregnant or lactating women
11. Women of childbearing potential (including women whose last menstrual period was less than one year prior to screening) who are unable or unwilling to use adequate contraception from study start to one year after the last dose of protocol therapy. Adequate contraception is defined as hormonal birth control, intrauterine device, double barrier method or total abstinence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2013-12; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
• The proportion of patients who can first de-escalate their treatment (to half the standard dose of their TKI) for 12 months, and then stop treatment completely for a further 2 years, without losing MMR. | 37months
  • The proportion of patients who can first de-escalate their treatment (to half the standard dose of their TKI) for 12 months, and then stop treatment completely for a further 2 years, without losing MMR.

SECONDARY OUTCOMES:
• Proportion of patients who can successfully de-escalate their treatment (to half the standard dose of their TKI), but who then lose MMR on complete TKI cessation | 37 months
  • Proportion of patients who can successfully de-escalate their treatment (to half the standard dose of their TKI), but who then lose MMR on complete TKI cessation
• Proportion of patients who lose their MMR on de-escalation/stopping and regain MMR on resumption of their TKI | 37 months
  • Proportion of patients who lose their MMR on de-escalation/stopping and regain MMR on resumption of their TKI
• Quality of Life | 37 months
  • Quality of Life
• Health Economic Assessment | 37 months
  • Health Economic Assessment
• Lab studies to define subsets of patients who are more likely to relapse on de-escalation / cessation. | 37 months
  • Lab studies to define subsets of patients who are more likely to relapse on de-escalation / cessation.

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Clark, MA MD, Principal Investigator — University of Liverpool
Locations (1):
- University of Liveprool, Liverpool, United Kingdom

REFERENCES:
- [Derived] Clark RE, Polydoros F, Apperley JF, Milojkovic D, Rothwell K, Pocock C, Byrne J, de Lavallade H, Osborne W, Robinson L, O'Brien SG, Read L, Foroni L, Copland M. De-escalation of tyrosine kinase inhibitor therapy before complete treatment discontinuation in patients with chronic myeloid leukaemia (DESTINY): a non-randomised, phase 2 trial. Lancet Haematol. 2019 Jul;6(7):e375-e383. doi: 10.1016/S2352-3026(19)30094-8. Epub 2019 Jun 12. PMID 31201085
- [Derived] Clark RE, Polydoros F, Apperley JF, Milojkovic D, Pocock C, Smith G, Byrne JL, de Lavallade H, O'Brien SG, Coffey T, Foroni L, Copland M. De-escalation of tyrosine kinase inhibitor dose in patients with chronic myeloid leukaemia with stable major molecular response (DESTINY): an interim analysis of a non-randomised, phase 2 trial. Lancet Haematol. 2017 Jul;4(7):e310-e316. doi: 10.1016/S2352-3026(17)30066-2. Epub 2017 May 26. PMID 28566209
- See also: Related Info — http://lctu.org.uk

DOCUMENTS (2):
  • Study Protocol (2018-05-24): https://cdn.clinicaltrials.gov/large-docs/85/NCT01804985/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-17): https://cdn.clinicaltrials.gov/large-docs/85/NCT01804985/SAP_001.pdf